CLINICAL TRIAL: NCT03499509
Title: Obesity Risk in African American Women is Determined by a Diet-by-phenotype Interaction
Acronym: CHAMPION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara Gower, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001324; R01DK115483-01A1 (NIH)
Record Dates: First submitted 2018-04-04; First posted 2018-04-17 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Diet Modification
MeSH Terms: interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Diet (Experimental): Low Glycemic (LG) diet: The LG diet was made up of foods that do not stimulate insulin secretion and was composed of 20% CHO, 55% fat, and 25% protein. The diet emphasized complex over simple carbohydrates and allowed dairy products, fruits, and vegetables within allowance of the diet.
  Interventions: Other: Low Glycemic Diet
- High Glycemic Diet (Placebo Comparator): High Glycemic (HG) diet: The HG diet aligned with the United States Department of Agriculture (USDA) guidelines (http://health.gov/dietaryguidelines/2015/guidelines/) and was composed of 55% CHO, 20% fat, and 25% protein. The diet emphasized complex over simple carbohydrates and allowed dairy products, fruits, and vegetables within allowance of the diet.
  Interventions: Other: High Glycemic Diet

INTERVENTIONS:
Other: Low Glycemic Diet — Low Glycemic (LG) diet: The LG diet was made up of foods that do not stimulate insulin secretion and was composed of 20% CHO, 55% fat, and 25% protein. The diet emphasized complex over simple carbohydrates and allowed dairy products, fruits, and vegetables within allowance of the diet.
  Other Names: Low Carbohydrate Diet
  Arms: Low Glycemic Diet
Other: High Glycemic Diet — High Glycemic (HG) diet: The HG diet aligned with the United States Department of Agriculture (USDA) guidelines (http://health.gov/dietaryguidelines/2015/guidelines/) and was composed of 55% CHO, 20% fat, and 25% protein. The diet emphasized complex over simple carbohydrates and allowed dairy products, fruits, and vegetables within allowance of the diet.
  Other Names: Low Fat Diet
  Arms: High Glycemic Diet

SUMMARY:
The Scientific Premise of this study is that the high level of obesity displayed by African American (AA) women is due to the ability to secrete large amounts of insulin when sugary foods are consumed. When AA women eat a diet rich in starchy or sugary food (a "high-glycemic" diet that stimulates insulin secretion), the food that is eaten is stored as fat rather than being burned as fuel. The investigators previous research has suggested that AA women have an easier time losing weight and keeping it off when eating a low-glycemic diet. The proposed study will be the first randomized clinical trial to test the effect of high and low glycemic diets for weight loss and weight-loss-maintenance in obese AA women.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-45 kg/m2
* Sedentary to moderately active (<2 hours/wk of moderate, structured, intentional exercise.
* Normal menstrual cycle

Exclusion Criteria:

* History of eating disorder
* daily use of tobacco (>1 pack/wk)
* change in weight greater than 5 pounds in previous 3 months
* presence of any condition (e.g. PCOS) or use of any medication (e.g. glucocorticoid) deemed by the project physician to interfere with study outcomes
* applicants will be screened with a standard oral glucose tolerance test. If a participant's 2 hour glucose if >200, they will not be able to enroll in the study.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gower, PhD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Lopez Torres SY, Gower BA, Garvey WT, Martins C. Adaptive Thermogenesis After Hypocaloric Low-Carbohydrate Versus Low-Fat Diets in African American Women: A Secondary Analysis. Obesity (Silver Spring). 2025 Nov;33(11):2160-2169. doi: 10.1002/oby.70020. Epub 2025 Sep 10. PMID 40931394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Glycemic Diet | High Glycemic Diet
Started | 34 | 33
Completed | 23 | 21
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Glycemic Diet | High Glycemic Diet | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 33 | 67
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Energy Expenditure
Description: Total energy expenditure measured by doubly labeled water. The protocol is based on established procedures [12]. Urine samples are analyzed in duplicate for H218O and 2H2O enrichments using Thermo Scientific Delta V Advantage IRMS with GasBench. CO2 production rates are determined using a fixed assumption for the dilution space ratio (1.043), using Equation 3 of Speakman et al. [10], and energy expenditure is calculated with equation 5 of Speakman et al. [10].
  [10] Speakman JR, Yamada Y, Sagayama H et al. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med 2021; 2:100203.
  [12] Goran MI, Carpenter WH, McGloin A et al. Energy expenditure in children of lean and obese parents. American Journal of Physiology 1995; 31:E917-E924.
  [13] Wolfe RR. Measurement of Total Energy Expenditure Using the Doubly-Labeled Water Method. In: Radioactive and Stable Isotope Tracers in Biomedicine. Edited by: Wiley-Liss. 1992.
Time Frame: Baseline, Week 13
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Low Glycemic Diet | High Glycemic Diet
Number analyzed (Participants) | 23 | 21
kcal/day
  Baseline | 2411 (342) | 2316 (289)
  week 13 | 2318 (362) | 2179 (413)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Low Glycemic Diet | High Glycemic Diet
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03499509/Prot_SAP_000.pdf